CLINICAL TRIAL: NCT06851507
Title: A Pilot Clinical Trial Comparing Topical Fluorouracil to Fluorouracil Plus Calcipotriene Field Treatments in Patients With Multiple Actinic Keratoses
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2003; NCI-2025-01497 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Multiple Actinic Keratoses
MeSH Terms: interventions — Fluorouracil; calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Fluorouracil and Calcipotriene (Experimental): Participants will screened and enrolled during a standard-of-care clinical dermatology visit. Participants will be randomized in between treatment with topical 5-FU twice daily for 2-3 weeks
  Interventions: Drug: Fluorouracil/Calcipotriene
- Treatment with Fluorouracil (Experimental): Participants will screened and enrolled during a standard-of-care clinical dermatology visit. Participants will be randomized in between treatment with topical 5-FU twice daily for 2-3 weeks
  Interventions: Drug: Fluorouracil 5-FU

INTERVENTIONS:
Drug: Fluorouracil 5-FU — Participants in the fluorouracil arm will apply fluorouracil twice daily for 2-3 weeks (depending on body area).
  Arms: Treatment with Fluorouracil
Drug: Fluorouracil/Calcipotriene — Participants in the fluorouracil/calcipotriene will apply fluorouracil/calcipotriene twice daily for 4 days to the affected area.
  Arms: Treatment with Fluorouracil and Calcipotriene

SUMMARY:
The goal of this clinical research study is to compare the effects of topical fluorouracil alone to topical fluorouracil plus topical calcipotriene in patients with multiple actinic keratoses. "Topical" means the medication is applied directly to the skin.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective of this pilot trial is feasibility, specifically measured by percent of patients approached and screened who enroll in the study. The prior trial on these medications reported a 75% enrollment rate (132 enrolled of 175 patients screened), though other trials of AK treatments have had lower enrollment rates (e.g., 53%9). To accurately plan a multi-site trial and apply for funding, an enrollment rate from the pilot trial will be critical. We will consider 50% enrollment rate a success, based on the lowest enrollment rates we found in the AK trial literature.

Secondary Objectives:

A. The proportion of participants who complete the treatment course, B. The change in AK count from baseline C. The proportion of participants who have clearance of >75% of AKs D. Differences in adverse event reporting, in particular redness, scaling, burning, pain, and itch, E. Comparison of counts of AK lesions by dermatologists in person to counts of AK lesions by dermatologists using standardized digital photography.

F. Change in MASCK metric G. Patient satisfaction (AK-EPQ) H. Change in health related QoL (AK-QoL) I. Patient adherence (ability to complete entire recommended course)

ELIGIBILITY:
Inclusion Criteria:

* Ability to start treatment within 1 week of enrollment
* Patients must be age ≥18, not of childbearing potential, and have the presence of 4-15 clinically, visibly confirmed and discrete AKs in an at least 25 cm2 contiguous area on the head, neck, arm, or hand.

Because no dosing or adverse event data are currently available on the use of fluorouracil in combination with calcipotriene in patients <18 years of age, children are excluded from this study.

* Patients with a prior or concurrent malignancy whose natural history or treatment does not interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* The effects of topical fluorouracil and/or fluorouracil plus calcipotriene on the developing human fetus are unknown. From the topical fluorouracil package insert: "One birth defect (cleft lip and palate) has been reported in the newborn of a patient using EFUDEX as recommended. One birth defect (ventricular septal defect) and cases of miscarriage have been reported when EFUDEX was applied to mucous membrane areas. Multiple birth defects have been reported in a fetus of a patient treated with intravenous fluorouracil."11 For this reason, we are excluding women of child-bearing potential. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

Postmenopausal (no menses in greater than or equal to 12 consecutive months). History of hysterectomy or bilateral salpingo-oophorectomy. Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).

History of bilateral tubal ligation or another surgical sterilization procedure.

• Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Known allergy to any component of the medications or vehicle.
* A wound or suspected skin cancer within 5cm of the area to be treated
* Immunosuppression, or use in the past month of medications that could impede skin assessment including but not limited to:

Other topical medications with active ingredients including: topical steroids, topical calcineurin inhibitors, topical retinoids, imiquimod, diclofenac, etc.

Artificial tanners Cytotoxic medications including: systemic fluorouracil, bleomycin, doxorubicin, cisplatin, etc.

Ultraviolet therapy Oral nicotinamide Oral retinoids including: isotretinoin, acitretin

* History of hypercalcemia
* Clinical evidence of vitamin D toxicity
* The effects of topical fluorouracil and/or fluorouracil plus calcipotriene on the developing human fetus are unknown. From the topical fluorouracil package insert: "One birth defect (cleft lip and palate) has been reported in the newborn of a patient using EFUDEX as recommended. One birth defect (ventricular septal defect) and cases of miscarriage have been reported when EFUDEX was applied to mucous membrane areas. Multiple birth defects have been reported in a fetus of a patient treated with intravenous fluorouracil."11 For this reason, we are excluding women of child-bearing potential. This includes all female patients, between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following:

Postmenopausal (no menses in greater than or equal to 12 consecutive months). History of hysterectomy or bilateral salpingo-oophorectomy. Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).

History of bilateral tubal ligation or another surgical sterilization procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mackenzie Wehner, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org